CLINICAL TRIAL: NCT02008331
Title: EFFECT OF SHORT-TERM TREATMENT WITH THE SYNBIOTIC PROBINUL-NEUTRO® ON GASTROINTESTINAL SYMPTOMS AND CIRCULATING PLASMA p-CRESOL LEVEL IN PATIENTS WITH CHRONIC RENAL FAILURE: A RANDOMIZED DOUBLE BLIND PILOT STUDY.
Brief Title: Effect of the Synbiotic Probinul-Neutro® on Gastrointestinal Symptoms and Plasma p-Cresol Level in Chronic Renal Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Bruna Guida, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Guida56
Record Dates: First submitted 2013-12-02; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; p-cresol; synbiotic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SYNBIOTIC (Experimental): Patients of this group assumed Probinul-Neutro® po 5g three times a day for 30 days
  Interventions: Dietary Supplement: SYNBIOTIC
- PLACEBO (Placebo Comparator): patients of this group received 5g of placebo 3 times a day for 30 days

INTERVENTIONS:
Dietary Supplement: SYNBIOTIC — INTERVENTION: Probinul neutro® assumed three times a day far from meals as 5 g powder packets dissolved in water. Probinul neutro® contains 5×109 Lactobacillus plantarum, 2×109 Lactobacillus casei subp. rhamnosus and 2×109 Lactobacillus gasseri, 1×109 Bifidobacterium infantis and 1×109 Bifidobacterium longum, 1×109 Lactobacillus acidophilus, 1×109 Lactobacillus salivarus and 1×109 Lactobacillus sporogenes and 5×109 Streptococcus termophilus, prebiotic inulin (2.2 g; VB Beneo Synergy 1) and 1.3 g of tapioca-resistant starch.
  PLACEBO: Tapioca-resistant starch powder similar in colour, texture and taste to the symbiotic mixture, assumed three times a day far from meals as 5 g powder packets dissolved in water.
  Other Names: Probinul-Neutro® or PLACEBO
  Arms: SYNBIOTIC

SUMMARY:
The interest on gastrointestinal (GI) dysfunction in CKD has been growing in the last years. it is now accepted that GI dysfunction in dialyzed patients may contribute to systemic microinflammation by promoting gut dysbiosis and bacterial translocation in the blood. Another mechanism by which GI dysfunction contributes to systemic symptoms in CKD is related to metabolic activity of the dysbiotic microflora growing in the gut of these patients to generate toxic compounds such as phenols, indoles, and amines. Epidemiological evidence has strongly linked one of these compounds, p-Cresol, to cardiovascular risk and mortality in CKD. In the present paper the investigators investigated the effect of a probiotic/prebiotic mixture on plasma p-cresol concentrations and GI symptoms and in CKD patients not on dialysis yet.

DETAILED DESCRIPTION:
In patients with chronic kidney disease (CKD), alterations in gut microbioma are posited to be responsible for gastrointestinal symptoms and generation of p-cresol, a uremic toxin, that has been associated to CKD progression and cardiovascular mortality.

This double blind randomized placebo controlled pilot study evaluates whether Probinul-neutro®, a synbiotic preparation that normalizes intestinal microflora, may lower plasma p-cresol concentrations and reduce gastrointestinal symptoms in non-dialyzed CKD patients.

Thirty patients on III-IV CKD stages were randomized to receive either Probinul neutro® or placebo for four weeks. Total plasma p-cresol concentrations was assessed at baseline, and 15 and 30 days after treatment start. At the same study times, ease and frequency of defecation, upper and lower abdominal pain, stool shape, borborygmi and flatus were quantified by subjective assessment questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* eGFR between 20 and 60 mL/min (stage 3-4 CKD, according to the K/DOQI CKD classification)

Exclusion Criteria:

* severe infections
* diabetes
* malignancy
* history of food intolerance
* autoimmune disorders
* severe malnutrition
* clinical conditions requiring artificial feeding
* kidney transplant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes in plasma p-cresol concentration | 30 days
  Fasting blood samples were drawn for the p-cresol plasma level

SECONDARY OUTCOMES:
composite outcome of gastrointestinal symptoms | 30 days
  Patients were asked to fill in a form for the scored evaluation of gastrointestinal symptoms (upper and inferior abdominal pain, borborygmus and flatus defecation frequency or easeand stool), and stool shape (Bristol stool chart)

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Guida, MD, Principal Investigator — Federico II University of Naples, ITALY
Locations (1):
- Federico II University of Naples, Naples, Naples, Italy

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148
- [Derived] Guida B, Germano R, Trio R, Russo D, Memoli B, Grumetto L, Barbato F, Cataldi M. Effect of short-term synbiotic treatment on plasma p-cresol levels in patients with chronic renal failure: a randomized clinical trial. Nutr Metab Cardiovasc Dis. 2014 Sep;24(9):1043-9. doi: 10.1016/j.numecd.2014.04.007. Epub 2014 May 2. PMID 24929795